CLINICAL TRIAL: NCT06133361
Title: Evaluation of the Rate and Type of Orthodontic Tooth Movement When Injecting Platelet-rich Plasma During Mini-implant-based Segmented En-masse Retraction of Upper Anterior Teeth: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Platelet-rich Plasma on the Rate and Type of Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-13-2023
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental): PRP will be injected in the palatal mucosa of the upper anterior teeth to accelerate orthodontic tooth movement. Patients in this group will undergo en-masse retraction of their upper front teeth using the same technique as the control group.
  Interventions: Biological: PRP injection
- Traditional retraction group (Active Comparator): In this group, patients will undergo en-masse retraction of their upper front teeth using a frictionless method by using coil springs attached between the anterior portion of the dental arch (which is an anterior segment only) to the miniscrews placed between the upper second premolars and the upper first molars.
  Interventions: Procedure: En-masse retraction of upper anterior teeth

INTERVENTIONS:
Biological: PRP injection — The PRP will be prepared according to a well-established technique and then injected into the palatal mucosa of the upper anterior teeth before retraction.
  Other Names: platelet-rich plasma (PRP)
  Arms: PRP group
Procedure: En-masse retraction of upper anterior teeth — The anterior teeth will be moved backward in an en-masse retraction way using a frictionless method. The anterior teeth will be manipulated as one block. Coil springs will be stretched between the power arms (in the anterior area) to the miniscrews placed in the posterior area bilaterally.
  Arms: Traditional retraction group

SUMMARY:
This study aims to assess the effect of PRP on the rate and type of OTM during en-masse frictionless retraction of maxillary anterior teeth using a segmental arch technique.

Thirty adult patients exhibiting class II division 1 malocclusion requiring upper first premolar extractions followed by en-masse retraction will participate in the study. They will be randomly and equally distributed into the PRP group (G1) and the control group (G2). The injection of PRP will be performed pre-retraction. The rate of orthodontic tooth movement will be assessed clinically by measuring the extraction space with a digital caliper. The cephalometric radiographs will evaluate the type of OTM at the beginning of en-masse retraction (T0) and at the middle of en-masse retraction (T1).

DETAILED DESCRIPTION:
One of the most important challenges in daily practice is prolonged orthodontic treatment duration. Many therapeutic procedures, such as chemical interventions, have been introduced to minimize orthodontic treatment time. Even though all the methods of chemically assisted acceleration of OTM increase the rate of bone turnover and increase the rate of tooth movement, however, these chemical agents, i.e., hormones or vitamin D3, have many problems such as systemic effects and short half-life which make them not practical in clinical orthodontic. Therefore, the injection of PRP has been proposed.

-In both groups, two first upper premolars were extracted. In all patients, fixed metal orthodontic brackets with MBT prescription 0.022 were bonded. After the arches were leveled and aligned, a rigid sectional archwire (0.021 x 0.025 in stainless steel) was used for the anterior six teeth. To strengthen anchorage, microscrews (diameter 1.6 mm; length 10 mm) were inserted at 8mm from the archwire into the inter-radicular space between the maxillary first molar and second premolar.

Two crimpable hooks were used with a height of 8 mm between the lateral incisor and canine on both sides of the sectional wire 0.021x0.025 to pass the force vector as close as possible to the center of resistance. En-masse retraction began one week after premolar extraction, using calibrated nickel-titanium coil springs with 175 g force per side.

-In PRP, 48 ml of blood was collected from the patient in sterile tubes with ACD-A as an anticoagulant. PRP was prepared as follows: Initially, the blood was centrifuged at 2000 rpm for 6 minutes. After separation of the blood, PRP and some Platelet-Poor Plasma (PPP) were collected and mixed in a dry tube, and then a second centrifugation was done at 2700 rpm for 3 minutes. After the second centrifugation, the lower 1/3rd of the tube is PRP. About 4 ml of PRP was collected from the tube, and then the patient was injected with it. After regional anesthesia for pain control, 0.5 ml of PRP was slowly injected submucosally palatal to each tooth from the right canine to the left canine using a 1cc syringe. Paracetamol was described for the patient to control pain and ensure confirming not to use ibuprofen or another NSAIDS. The injection was applied one time.

ELIGIBILITY:
Inclusion Criteria:

1. age range between 16 and 27 years
2. Class II division I malocclusion in which extraction of upper first premolars is indicated
3. skeletal class II relationships (4°<ANB<10°),
4. Non-growing patients
5. No maxillary constriction
6. overjet >5 and <10 mm
7. normal overbite of 0-50%
8. normal anterior facial height
9. No systemic disease.

Exclusion Criteria:

1. patients who have undergone previous orthodontic treatment
2. patients who need orthopedic surgery
3. moderate to severe anterior crowding (Disharmony Dento-Maxillary (DDM≥3)
4. Poor oral hygiene,
5. long-term use of medical drugs, especially NSAIDs

Ages: 16 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-24 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Rate of retraction | At the middle of the retraction procedure (the middle of closing the extraction space); this assessment time is expected to occur within 2 to 3 months and 3 to 4 months after the onset of retraction in the experimental and control groups, respectively
  Assessment will be performed clinically by measuring the change in the extraction space. The amount of distance being retracted in millimeters will be divided by the duration of retraction in months to estimate the retraction rate.
Change in incisors' positions | First time point (T0): one day before the beginning of retraction. Second time point (T1): in the middle of extraction space closure (expected to be within 2-3 months in the exp. group and 3-4 months in the control group).
  The position of the incisal edges of the upper incisors will be measured according to a reference plance.
Change in position of the root apex of the incisor vertically (UIA-v). | First time point (T0): one day before the beginning of retraction. Second time point (T1): in the middle of extraction space closure (expected to be within 2-3 months in the exp. group and 3-4 months in the control group).
  This variable represents the distance between the upper root apex and X reference plane (line drawn from ANS to PNS which is called the palatal plane SPP). Lateral cephalograms will be taken, and this variable will be measured in millimeters.
Change in position of the incisal edge of the incisor vertically (UIE-v). | First time point (T0): one day before the beginning of retraction. Second time point (T1): in the middle of extraction space closure (expected to be within 2-3 months in the exp. group and 3-4 months in the control group).
  This variable represents the distance between the upper incisal edge and X reference plane. Lateral cephalograms will be taken and this variable is going to be measured in millimeters.
Change in position of the root apex of the incisor horizontally (UIA-h) | First time point (T0): one day before the beginning of retraction. Second time point (T1): in the middle of extraction space closure (expected to be within 2-3 months in the exp. group and 3-4 months in the control group).
  This variable represents the distance between the upper root apex and Y reference plane (line perpendicular to SPP at lateral PT). Lateral cephalograms will be taken and this variable is going to be measured in millimeters.
Change in position of the incisal edge of the incisor horizontally (UIE-h) | First time point (T0): one day before the beginning of retraction. Second time point (T1): in the middle of extraction space closure (expected to be within 2-3 months in the exp. group and 3-4 months in the control group).
  This variable represents the distance between the upper incisal edge and Y reference line. Lateral cephalograms will be taken and this variable is going to be measured in millimeters.

SECONDARY OUTCOMES:
Change in the UI/SPP angle | First time point (T0): one day before the beginning of retraction. Second time point (T1): in the middle of extraction space closure (expected to be within 2-3 months in the exp. group and 3-4 months in the control group).
  This angle represents the inclination of the upper incisors (UI) relative to the palatal plane (or spinal plane SPP) in the sagittal direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the SNA angle | First time point (T0): one day before the beginning of retraction. Second time point (T1): in the middle of extraction space closure (expected to be within 2-3 months in the exp. group and 3-4 months in the control group).
  This angle represents the position of the upper jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in the ANB angle | First time point (T0): one day before the beginning of retraction. Second time point (T1): in the middle of extraction space closure (expected to be within 2-3 months in the exp. group and 3-4 months in the control group).
  This angle represents the spatial relationship between the upper and lower jaws in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken, and this angle will be measured in degrees.
Change in Overbite | First time point (T0): one day before the beginning of retraction. Second time point (T1): in the middle of extraction space closure (expected to be within 2-3 months in the exp. group and 3-4 months in the control group).
  This variable represents The vertical overlap of the maxillary incisors over the mandibular incisors, measured relative to the incisal edges. Lateral cephalograms will be taken, and this variable will be measured in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Y Hajeer, DDS MSc PhD, Study Director — Professor of Orthodontics, Department of Orthodontics, Faculty of Dentistry, University of Damascus
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, Aleppo University, Aleppo, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khlef HN, Hajeer MY, Ajaj MA, Heshmeh O. Evaluation of Treatment Outcomes of En masse Retraction with Temporary Skeletal Anchorage Devices in Comparison with Two-step Retraction with Conventional Anchorage in Patients with Dentoalveolar Protrusion: A Systematic Review and Meta-analysis. Contemp Clin Dent. 2018 Oct-Dec;9(4):513-523. doi: 10.4103/ccd.ccd_661_18. PMID 31772456
- [Background] Ozaki H, Tominaga JY, Hamanaka R, Sumi M, Chiang PC, Tanaka M, Koga Y, Yoshida N. Biomechanical aspects of segmented arch mechanics combined with power arm for controlled anterior tooth movement: A three-dimensional finite element study. J Dent Biomech. 2015 Jan 8;6:1758736014566337. doi: 10.1177/1758736014566337. eCollection 2015. PMID 25610497
- [Background] Al-Naoum F, Hajeer MY, Al-Jundi A. Does alveolar corticotomy accelerate orthodontic tooth movement when retracting upper canines? A split-mouth design randomized controlled trial. J Oral Maxillofac Surg. 2014 Oct;72(10):1880-9. doi: 10.1016/j.joms.2014.05.003. Epub 2014 May 14. PMID 25128922
- [Background] Al-Imam GMF, Ajaj MA, Hajeer MY, Al-Mdalal Y, Almashaal E. Evaluation of the effectiveness of piezocision-assisted flapless corticotomy in the retraction of four upper incisors: A randomized controlled clinical trial. Dent Med Probl. 2019 Oct-Dec;56(4):385-394. doi: 10.17219/dmp/110432. PMID 31794163
- [Background] Gulec A, Bakkalbasi BC, Cumbul A, Uslu U, Alev B, Yarat A. Effects of local platelet-rich plasma injection on the rate of orthodontic tooth movement in a rat model: A histomorphometric study. Am J Orthod Dentofacial Orthop. 2017 Jan;151(1):92-104. doi: 10.1016/j.ajodo.2016.05.016. PMID 28024792
- [Background] Angel SL, Samrit VD, Kharbanda OP, Duggal R, Kumar V, Chauhan SS, Coshic P. Effects of submucosally administered platelet-rich plasma on the rate of tooth movement. Angle Orthod. 2022 Jan 1;92(1):73-79. doi: 10.2319/011221-40.1. PMID 34491291
- [Background] Al-Sibaie S, Hajeer MY. Assessment of changes following en-masse retraction with mini-implants anchorage compared to two-step retraction with conventional anchorage in patients with class II division 1 malocclusion: a randomized controlled trial. Eur J Orthod. 2014 Jun;36(3):275-83. doi: 10.1093/ejo/cjt046. Epub 2013 Jun 20. PMID 23787192